CLINICAL TRIAL: NCT00692120
Title: Clinical Approaches to Correcting Vitamin D Inadequacy and Maintaining Adequacy
Acronym: D2/D3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-0013
Record Dates: First submitted 2008-01-02; First posted 2008-06-06 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-04

CONDITIONS: Vitamin D Inadequacy; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Dietary Supplement: Ergocalciferol (vitamin D2); Dietary Supplement: Placebo
- 2 (Experimental)
  Interventions: Dietary Supplement: Ergocalciferol (vitamin D2); Dietary Supplement: Placebo
- 3 (Experimental)
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3); Dietary Supplement: Placebo
- 4 (Experimental)
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3); Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (vitamin D3) — 50,000 IU once monthly for 12 months
  Arms: 3
Dietary Supplement: Ergocalciferol (vitamin D2) — oral capsule 50,000 IU once monthly for 12 months
  Arms: 1
Dietary Supplement: Ergocalciferol (vitamin D2) — oral capsule 1600 IU once daily for 12 months
  Arms: 2
Dietary Supplement: Cholecalciferol (vitamin D3) — oral capsule 1600 IU once daily for 12 months
  Arms: 4
Dietary Supplement: Placebo — oral placebo capsule once daily for 12 months

SUMMARY:
Vitamin D is available in two forms, vitamin D2 and vitamin D3. It has previously been assumed that these two forms maintain blood vitamin D equally. However, this may not be the case. This study will evaluate whether D2 and D3 produce equal elevation of blood vitamin D. Additionally, it will evaluate whether once per month vitamin D dosing is as effective in maintaining blood vitamin D levels as daily dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Community dwelling men and women age ≥ 65 years.
2. Able and willing to sign informed consent.
3. Serum 25OHD concentration ≥ 10 and less than 60 ng/ml by HPLC.
4. Willing to avoid use of cod-liver oil and non-study vitamin D supplementation; standard multiple vitamins containing ≤ 400 IU used no more than once daily will be allowed

Exclusion Criteria:

1. Current hypercalcemia (serum calcium > 10.5 mg/dl) or untreated primary hyperparathyroidism.
2. History of nephrolithiasis.
3. Screening 25OHD concentration ≥ 60 ng/ml.
4. Baseline 24-hour urine calcium > 250 mg if female, > 300 mg if male.
5. Known risk factors for hypercalcemia, e.g., malignancy, tuberculosis, sarcoidosis, Paget's disease
6. History of any form of cancer within the past five years with the exception of adequately treated squamous cell or basal cell skin cancer.
7. Renal failure defined as a calculated creatinine clearance (Cockroft-Gault method) ≤ 25 ml/minute
8. Severe end-organ disease, e.g., cardiovascular, hepatic, hematologic, pulmonary, etc., which may limit ability to complete the study
9. Known malabsorption syndromes, e.g., celiac disease, radiation enteritis, active inflammatory bowel disease, etc.
10. Use of medications known to alter bone turnover including bisphosphonates, estrogen, selective estrogen receptor modulators, PTH, testosterone or calcitonin
11. Vitamin D intake greater than 5,000 IU daily
12. Treatment with any active metabolites of vitamin D within six months of screening
13. Treatment with any drug which may interfere with vitamin D metabolism, e.g., phenobarbital, phenytoin.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is change in 25OHD with various D2 and D3 dosing regimens. | 12 months

SECONDARY OUTCOMES:
Determine whether once monthly vitamin D2 or D3 dosing is as effective as daily dosing in attainment, and subsequent maintenance, of 25OHD status | 12 months
Delineate the effect of these vitamin D regimens on other parameters of skeletal relevance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Principal Investigator — University of Wisconsin - Institute on Aging
Locations (1):
- UW Osteoporosis Clinical and Research Program, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Binkley N, Gemar D, Engelke J, Gangnon R, Ramamurthy R, Krueger D, Drezner MK. Evaluation of ergocalciferol or cholecalciferol dosing, 1,600 IU daily or 50,000 IU monthly in older adults. J Clin Endocrinol Metab. 2011 Apr;96(4):981-8. doi: 10.1210/jc.2010-0015. Epub 2011 Feb 2. PMID 21289249